CLINICAL TRIAL: NCT00937963
Title: Healthy FAT (Fatty Acids in Transition) Study
Brief Title: Healthy Fatty Acids in Transition
Acronym: FAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: California Healthcare Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PKE 103
Record Dates: First submitted 2009-06-18; First posted 2009-07-13 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: cholesterol; cardiovascular; CVD; Triglycerides; Heart
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palm Oil (Experimental): Traditional palm oil normally used in foods
  Interventions: Dietary Supplement: Palm DAG Oil

INTERVENTIONS:
Dietary Supplement: Palm DAG Oil — Use of Palm DAG Oil to replace palm oil traditionally used in foods

SUMMARY:
Diacylglycerol (DAG) is a molecule that consists of two fatty acid chains bound by ester links to a glycerol molecule, in the form of 1,2 and 1,3 structural isomers. Approximately 10% of the edible oils on today's market are comprised from DAG. DAG oil has a similar taste, appearance, and fatty acid composition as conventional triacylglycerol oil (TAG; consists of 3 fatty acids chains bound to a glycerol molecule), yet recent studies suggest that due to its different chemical structure, DAG oil may induce cardiovascular (CV) benefits. Specifically, human studies in the United States (US) and Japan have shown that long-term consumption of a diet containing DAG oil enhances loss of body weight and body fat compared with TAG oil of similar fatty acid composition. In postprandial studies, serum triglycerides (TG) and remnant like particle cholesterol concentrations, have shown to be lower following ingestion of DAG-enriched oil compared to conventional dietary oil (e.g., soybean, corn), or TAG oil. Therefore, DAG oil appears to be effective for preventing postprandial hyperlipidemia, which is a risk factor for arteriosclerosis.

The hypothesis that the investigators propose in this pilot study is that intake of DAG oil, compared to TAG oil will result in a lower LDL-C, and lower LDL-C/HDL-C ratio, as well as a reduction in TG levels. Given the significance of such findings, if confirmed, the investigators will evaluate other important clinical biomarkers for chronic disease (CV Disease, type 2 diabetes, metabolic syndrome), such as insulin sensitivity and inflammation [as determined by C-reactive protein (CRP), interleukin (IL)-1, IL-6 & tumor necrosis factor-alpha (TNF-α)], which also may be beneficially affected by consumption of the palm DAG oil. During the pilot study, the investigators will reserve serum/plasma samples so that these additional assays may be run upon approval of the modification.

DETAILED DESCRIPTION:
Commonly consumed vegetable fats and oils are comprised predominantly of TAG, and small amounts of DAG and monoacylglycerol. TAG consists of 3 fatty acid ester, whereas diacylglycerol oil has 2 fatty acid esters linked to a glycerol backbone. Recently, Watanabe et al., developed a process by which the ratio of glycerides found in plant oils such as soybean, canola (rapeseed), or corn can be shifted from TAG to DAG, leading to the formation of oil composed largely of DAG. Commercially, DAG oil is produced by esterification of fatty acids derived from natural edible plant oils in the presence of lipase enzyme. Commercially produced vegetable DAG oil contains >80% DAG, <20% TAG, <5% monoacylglycerols, and small amounts of emulsifiers and antioxidants to maintain quality. The main constituent fatty acids of DAG oil are oleic (C18:1), linoleic (C18:2), and linolenic (C18:3) acids, present as 1,3- and 1,2 (or 2,3)-DAGs in a ratio of 7:3, respectively. These structural differences may be responsible for the purported metabolic effects of DAG compared to TAG oil, DAG oil has fewer fatty acids than TAG, and DAG-oil with a greater proportion of DAG in the sn-1,3 versus sn-1,2 form may be more readily oxidized. Thus, the effects of DAG oil on increasing LDL-C would be expected to be less than TAG oil.

ELIGIBILITY:
Inclusion Criteria:

* 30-60 years of age
* Moderately elevated LDL-C (120-175 mg/dL) and normal HDL-C (30-50 mg/dL)
* TG < 350 mg/dL

Exclusion Criteria:

* Smokers
* A history of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease, and thyroid disease (unless controlled on medication)
* Lactation, pregnancy, or desire to become pregnant during the study
* Cholesterol-lowering medications
* Intake of putative cholesterol-lowering supplements (psyllium, fish oil capsules, soy lecithin, niacin, fiber, flax, and phytoestrogens, stanol/sterol supplemented foods)
* Vegetarianism
* Allergic to nuts (Other food allergies will be reviewed on a case-by-case basis)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Lipoprotein profile (total cholesterol, LDL-C, HDL-C, TG) | At the end of each 4 week diet period (week 4 and week 10)
  Participants receive a two week break between diet periods. Diet period 1 runs from week 1-4 and diet period 2 from week 7-10.

SECONDARY OUTCOMES:
Inflammatory markers (CRP, IL-1, IL-6 & TNF-α) | At the end of each 4 week diet period (week 4 and week 10)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States